CLINICAL TRIAL: NCT06808737
Title: Assessment of the Efficacy of Transversus Abdominis Plane Block in Alleviating Acute Appendicitis Pain in the Emergency Department
Brief Title: Efficacy of Transversus Abdominis Plane Block in Alleviating Acute Appendicitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AEŞH-EK1-2024-0038
Record Dates: First submitted 2024-08-14; First posted 2025-02-05 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-01

CONDITIONS: Acute Appendicitis
Keywords: Transversus Abdominis Plane block; Acute Appendicitis; Pain management; Emergency Department; Pain control; Analgesics, opioid; Bupivacaine; Analgesia
MeSH Terms: conditions — Appendicitis; Agnosia; Emergencies

STUDY DESIGN:
Intervention Model Description: The study will include patients who present to the emergency department with abdominal pain, receive a diagnosis of acute appendicitis through history, physical examination, and imaging modalities, and are determined to undergo definitive surgery following general surgical consultation. Patients will be randomly assigned to three groups.
Who Masked: Outcomes Assessor
Masking Description: The surgeon performing the surgery, the anesthesiologist, the nurses, and the emergency medicine doctor filling out the case form will be blinded to the patient groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- T-50 (No Intervention): Participants in the T-50 group will receive a 100 cc isotonic 0.9% NaCl (normal saline) solution containing 50 mg tramadol as an intravenous infusion over 15 minutes at baseline.
- TAP-50 (Active Comparator): Participants in the TAP-50 group will receive the same intravenous tramadol infusion as the T-50 group at baseline, followed by a transversus abdominis plane (TAP) block.
  Interventions: Procedure: Transversus Abdominis Plane Blockage
- TAP-100 (Active Comparator): Participants in the TAP-100 group will receive a 100 cc isotonic 0.9% NaCl solution containing 100 mg tramadol as an intravenous infusion over 15 minutes at baseline, followed by a TAP block.
  Interventions: Procedure: Transversus Abdominis Plane Blockage

INTERVENTIONS:
Procedure: Transversus Abdominis Plane Blockage — Patient monitoring will be conducted, followed by the preparation of the skin with 10% povidone-iodine and ensuring appropriate draping. A high-frequency linear transducer will be placed transversely between the right iliac crest and subcostal margin along the midaxillary line. Structures visualized on ultrasound from superficial to deep include: skin, subcutaneous fat, external oblique muscle, internal oblique muscle, transversus abdominis muscle, and peritoneum. The TAP block will be performed in the transversus abdominis plane (TAP) between the internal oblique and transversus abdominis muscles. A 23-gauge, 60 mm blunt-tipped needle will be directed toward the TAP, and negative aspiration will be confirmed upon entry into the fascial layer. An injection of 20 mL of 0.25% bupivacaine, prepared by diluting 10 mL of 0.5% bupivacaine with 10 mL of normal saline, will be performed, followed by the visualization of the oval spread of bupivacaine in the TAP.
  Arms: TAP-100; TAP-50

SUMMARY:
This study aims to evaluate the efficacy of Transversus Abdominis Plane (TAP) block in preoperative pain management for patients diagnosed with acute appendicitis who are scheduled for emergency surgery in the emergency department. The research seeks to assess the potential of TAP block in reducing pain intensity prior to surgical intervention among patients diagnosed with acute appendicitis in the emergency setting. The goal is to contribute insights that can enhance practical approaches to achieving optimal pain control for acute appendicitis patients in emergency department settings.

DETAILED DESCRIPTION:
This study will include patients who present to the emergency department with abdominal pain, receive a diagnosis of acute appendicitis through history, physical examination, and imaging modalities, and are determined to undergo definitive surgery following general surgical consultation. Participants will be randomly assigned to three groups. Randomization will be achieved by allocating the first 5 patients to the T-50 group, the second 5 patients to the TAP-50 group, and the third 5 patients to the TAP-100 group. Following treatment, patients' Numeric Rating Scale (NRS) scores will be recorded at 30, 60, and 120 minutes during rest, coughing, and heel tap. If the NRS score is above 5, rescue analgesia will be administered as a 50 mcg fentanyl intravenous infusion over 15 minutes. Subsequently, patient demographic data including age, gender, height, weight, BMI, comorbidities, and medications, as well as vital signs upon admission, complete blood count values, coagulation parameters, creatine kinase levels, appendicitis rupture/non-rupture status, planned laparoscopic/open surgery, Alvarado score, time to first rescue analgesia after baseline analgesia administration (minutes), total analgesic requirement in the emergency department (mg), and TAP block complications (hematoma, surgical site infection, intra-abdominal collection, intramuscular injection - myonecrosis) will be documented. Patient satisfaction will be assessed using a 5-point Likert scale. cutaneous sensory distribution will be assessed at 20 minutes following TAP block. Following this, operative duration (minutes), time to first rescue analgesia postoperatively (minutes), postoperative 2, 4, 6, 12, 24-hour nausea-vomiting (PONV) score, NRS scores during rest, coughing, and heel tap at postoperative 2, 4, 6, 12, 24 hours, cumulative analgesic medications at postoperative 2, 4, 6, 12, 24 hours, postoperative rescue antiemetic requirement, total analgesic cost, and length of hospital stay (days) will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with acute appendicitis in the emergency department and scheduled for definitive surgery following general surgical consultation: patients will have their Alvarado score calculated based on history, physical examination, and laboratory tests, and acute appendicitis will be confirmed by ultrasound and/or contrast-enhanced/non-contrast-enhanced abdominal CT.
* Patients aged 18 and over
* Patients who provide written consent

Exclusion Criteria:

* Patients with abdominal wall anatomical abnormalities
* Patients with known local anesthetic allergies
* Body mass index > 30
* Patients weighing less than 45 kg
* Coagulopathy
* Patients with opioid, alcohol, or substance addiction
* Patients with skin infections at the site of local anesthetic application
* Pregnant or breastfeeding patients
* Hemodynamically unstable patients
* Patients with liver or kidney failure
* Patients with chronic pain disorders
* Patients who have difficulty cooperating or have language barriers
* Patients who do not provide written consent
* Patients under 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2024-05-08 (Actual); Primary Completion 2025-05-08 (Estimated); Study Completion 2025-05-09 (Estimated)

PRIMARY OUTCOMES:
Need for opioids (mg) for effective pain relief according to NRS | Approximately 1 year after study start date
  Determination of whether TAP block reduces the need for opioids in the management of acute appendicitis pain in the emergency department.

SECONDARY OUTCOMES:
Pain assessed by NRS | Approximately 1 year after study start date
  Evaluation of the effectiveness of multimodal pain control for acute appendicitis pain in the emergency department across different groups.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmet Burak Erdem, Assoc. Prof., Principal Investigator — Ankara Etlik City Hospital
Locations (1):
- Ankara City Hospital, Ankara, Yenimahalle, Turkey (Türkiye)

REFERENCES:
- [Background] Scholl L, Seth P, Kariisa M, Wilson N, Baldwin G. Drug and Opioid-Involved Overdose Deaths - United States, 2013-2017. MMWR Morb Mortal Wkly Rep. 2018 Jan 4;67(5152):1419-1427. doi: 10.15585/mmwr.mm675152e1. PMID 30605448
- [Background] Falch C, Vicente D, Haberle H, Kirschniak A, Muller S, Nissan A, Brucher BL. Treatment of acute abdominal pain in the emergency room: a systematic review of the literature. Eur J Pain. 2014 Aug;18(7):902-13. doi: 10.1002/j.1532-2149.2014.00456.x. Epub 2014 Jan 22. PMID 24449533
- [Background] Freys JC, Bigalke SM, Mertes M, Lobo DN, Pogatzki-Zahn EM, Freys SM; PROSPECT Working Group of the European Society of Regional Anaesthesia and Pain Therapy (ESRA). Perioperative pain management for appendicectomy: A systematic review and Procedure-specific Postoperative Pain Management recommendations. Eur J Anaesthesiol. 2024 Mar 1;41(3):174-187. doi: 10.1097/EJA.0000000000001953. Epub 2024 Jan 12. PMID 38214556
- [Background] Tsai HC, Yoshida T, Chuang TY, Yang SF, Chang CC, Yao HY, Tai YT, Lin JA, Chen KY. Transversus Abdominis Plane Block: An Updated Review of Anatomy and Techniques. Biomed Res Int. 2017;2017:8284363. doi: 10.1155/2017/8284363. Epub 2017 Oct 31. PMID 29226150
- [Result] Chou R, Gordon DB, de Leon-Casasola OA, Rosenberg JM, Bickler S, Brennan T, Carter T, Cassidy CL, Chittenden EH, Degenhardt E, Griffith S, Manworren R, McCarberg B, Montgomery R, Murphy J, Perkal MF, Suresh S, Sluka K, Strassels S, Thirlby R, Viscusi E, Walco GA, Warner L, Weisman SJ, Wu CL. Management of Postoperative Pain: A Clinical Practice Guideline From the American Pain Society, the American Society of Regional Anesthesia and Pain Medicine, and the American Society of Anesthesiologists' Committee on Regional Anesthesia, Executive Committee, and Administrative Council. J Pain. 2016 Feb;17(2):131-57. doi: 10.1016/j.jpain.2015.12.008. PMID 26827847